CLINICAL TRIAL: NCT06047145
Title: Evaluation of Oral Soy Isoflavone Concentrates on Skin Ageing Parameters: a Double-blind Randomised Placebo-controlled Trial
Brief Title: Evaluation of Soy Isoflavones on Skin Ageing Parameters
Acronym: ISOSKIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Archer-Daniels-Midland Company (Industry)
Collaborators: Eurofins Dermscan Pharmascan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CTB2022TN110
Record Dates: First submitted 2023-09-05; First posted 2023-09-21 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2024-03

CONDITIONS: Skin Ageing
Keywords: soy isoflavones; skin ageing; menopause
MeSH Terms: interventions — Soybean Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- soy isoflavones (Experimental): One oral capsule daily containing 200mg soy isoflavones for 84 days
  Interventions: Dietary Supplement: soy isoflavones
- placebo (Placebo Comparator): One oral capsule daily containing equivalent placebo for 84 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: soy isoflavones — 1 capsule daily for 84 days
  Arms: soy isoflavones
Dietary Supplement: Placebo — 1 capsule daily for 84 days
  Arms: placebo

SUMMARY:
This double-blind, placebo-controlled, randomised pilot trial aims to assess the effect of oral soy isoflavone consumption on skin ageing parameters in post-menopausal women.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subject.
2. Sex: female.
3. Age: from 40 to 65 years (inclusive).
4. Phototype: I to IV on the Fitzpatrick scale.
5. Post-menopausal subject, with last menstrual period at least 12 months prior to screening and who is not using hormonal contraception.
6. Subject having Crow's feet wrinkles from grade 2 to 5 on Bazin's scale.
7. Subject having under eyes wrinkles.
8. Subject agreeing not to change her alimentary and cosmetic habits during the study.
9. Subject, able to understand the study related information and to give a written informed consent.
10. Subject having given freely and expressly informed consent.
11. Subject able and willing to comply with protocol requirements.
12. Subject affiliated to a health social security system.

Exclusion Criteria:

1. Women with childbearing potential or women on long term hormonal contraception whose childbearing potential is difficult to ascertain.
2. Subject deprived of her freedom by administrative or legal decision.
3. Subject under guardianship or unable to provide consent.
4. Subject in a social or healthcare institution.
5. Subject suspected to be non-compliant according to the investigator's judgment.
6. Subject participating in any other clinical study or being in an exclusion period for a previous study.
7. Subject having crow's feet wrinkles with grades < 2 or > 5 on Bazin's scale.
8. Subject with a tattoo, a scar, moles, too many hairs or anything on the studied zones which might interfere with the evaluation.
9. Personal or family history of breast, uterine or ovarian cancer as per investigator judgement.
10. Subject with personal history of cancer.
11. Subject with a condition or receiving a medication which, in the investigator's judgement, put the subject at undue risk.
12. Subject suffering from a severe or progressive disease, likely to interfere with the measured parameters.
13. Subject with any skin or systemic disease (acute and/or chronic), ongoing or in the previous year, likely to interfere with the measured parameters or to put the subject at undue risk.
14. Subject with known history of or suffering from autoimmune disease and/or immune deficiency.
15. Subject with allergies or intolerance to soy or soy products.
16. Subject having history of allergy or hypersensitivity to any of the components of the tested product.
17. Subject under anti-coagulant treatment.
18. Subject under thyroid hormones treatment.
19. Subject under osteoporosis treatment other than vitamin D and calcium.
20. Subject having started or stopped supplements used to treat menopausal symptoms, which may affect measured parameters, such as phytoestrogens, Black Cohosh, dehydroepiandrosterone (DHEA), hyaluronic acid, collagen, NADH, resveratrol soy supplements, etc. within one month prior to screening.
21. Subject having received injection with botulinum toxin on Crow's feet wrinkles in the year before the screening visit.
22. Subject having received injection with botulinum toxin on other zone of the face in the past 6 months before the screening visit.
23. Subject having received injection of filling product on the studied zones (crow's feet and under eye wrinkles, cheekbones and forearms) in the year before the screening visit.
24. Subject having received tensor threads on the face in the two years before the screening visit.
25. Subject having received injection of mesotherapy in the face in the past 3 months before the screening visit.
26. Subject having received professional peeling on the face and forearms in the past 3 months before the screening visit.
27. Subject having received a treatment with a laser on the face or forearms in the past 6 months before the screening visit.
28. Subject under oral hormonal substitutive treatment during the year previous the screening visit.
29. Subject receiving any long-term medical treatment or any treatment that, in the opinion of the clinical investigator, may interfere with test results or put the subject at undue risk.
30. Subject undergoing a topical treatment on the test area (forearms and face) or a systemic treatment:

    * corticosteroids during the 2 previous weeks and during the study.
    * retinoids and/or immunosuppressors during the 3 previous months and during the study.
31. Intensive exposure to sunlight within the previous month and foreseen during the study without adequate sun protection, as per the investigator's judgement.
32. Exposure to artificial UV or spray tan in the month preceding the screening or during the study.
33. Subject with an excessive consumption of alcohol (more than 2 glasses of wine per day) and/or tobacco (more than 10 cigarettes per day).

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-10-27 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
Change in Crow's Feet wrinkles (Ra) | day 0, day 84
  Cutaneous relief parameters (Ra - Average roughness) on Crow's Feet wrinkles measured with fringe projection acquisitions

SECONDARY OUTCOMES:
Change in Crow's Feet wrinkles (Ra) | day 0, day 42
  Cutaneous relief parameters (Ra - Average roughness) on Crow's Feet wrinkles measured with fringe projection acquisitions
Change in Crow's Feet wrinkles (Rz) | day 0, day 42, day 84
  Cutaneous relief parameters (Rz - Average height of the roughness) on Crow's Feet wrinkles measured with fringe projection acquisitions
Change in Crow's Feet wrinkles (Rt) | day 0, day 42, day 84
  Cutaneous relief parameters (Rt - Maximum height of the roughness profile) on Crow's Feet wrinkles measured with fringe projection acquisitions
Change in under eye wrinkles (Ra) | day 0, day 42, day 84
  Cutaneous relief parameters (Ra - Average roughness) on under eye wrinkles measured with fringe projection acquisitions
Change in under eye wrinkles (Rt) | day 0, day 42, day 84
  Cutaneous relief parameters (Rt - Maximum height of the roughness profile) on under eye wrinkles measured with fringe projection acquisitions
Change in under eye wrinkles (Rz) | day 0, day 42, day 84
  Cutaneous relief parameters (Rz - Average height of the roughness) on under eye wrinkles measured with fringe projection acquisitions
Change in skin hydration | day 0, day 42, day 84
  Skin hydration will be evaluated by Corneometer® on the forearm.
Change in skin colour | day 0, day 42, day 84
  Skin colour will be evaluated by Spectrophotometer® on the cheekbone.
Change in skin barrier function | day 0, day 42, day 84
  Skin barrier function will be evaluated by the measurement of Trans Epidermal Water Loss with Aquaflux® on the forearm
Subject satisfaction | day 42, day 84
  A non-validated subjective evaluation questionnaire on the study product's effects on the skin will be completed by subjects (each item is scored individually on a 5 point Likert scale ranging from 'Totally agree' to 'Totally disagree')
Adverse events | day 0, day 42, day 84
  Collection of adverse events throughout the study

OTHER OUTCOMES:
Urinary isoflavones and metabolites | day 0, day 42, day 84
  To quantify levels of key isoflavones and metabolites in urine
Equol-producing status | day 0, day 42, day 84
  To identify equol-producing individuals based on urine levels of equol

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofins Dermscan Pharmascan, Villeurbanne, France

REFERENCES:
- [Derived] Vijayakumar V, Climent E, Enrique M, Lamelas A, Alvarez B, Chenoll E, Naghibi M, Day R. S-equol status modulates skin response to soy isoflavones in postmenopausal women: results from a randomized placebo-controlled pilot trial. Front Nutr. 2025 Nov 3;12:1671835. doi: 10.3389/fnut.2025.1671835. eCollection 2025. PMID 41256931